CLINICAL TRIAL: NCT01163838
Title: A Phase 1, Placebo-Controlled, Randomized Study To Assess The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Following Multiple Intravenous Doses Of RN316 In Healthy Adult Subjects With Hypercholesterolemia
Brief Title: Multiple-Dose Safety Study Of RN316 For TheTreatment Of Hypercholesterolemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was redesigned based on FDA feedback.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1481002
Record Dates: First submitted 2010-07-14; First posted 2010-07-16 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: Hypercholesterolemia; Dyslipidemia; LDL; Cholesterol; High Cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo
- RN316: 1 mg/kg every 2 weeks (Experimental)
  Interventions: Biological: 1 mg/kg every 2 weeks
- RN316: 2 mg/kg every 4 weeks (Experimental)
  Interventions: Biological: 2 mg/kg every 4 weeks
- RN316: 4 mg/kg every 4 weeks (Experimental)
  Interventions: Biological: 4 mg/kg every 4 weeks
- RN316: 4 mg/kg every 8 weeks (Experimental)
  Interventions: Biological: 4 mg/kg every 8 weeks
- RN316: 8 mg/kg every 8 weeks (Experimental)
  Interventions: Biological: 8 mg/kg every 8 weeks
- RN316: 12 mg/kg every 8 weeks (Experimental)
  Interventions: Biological: 12 mg/kg every 8 weeks

INTERVENTIONS:
Biological: Placebo — Subjects will receive placebo or active treatment every 2 weeks for a total of 9 doses. Duration of IV infusion is 60 minutes. Total dose is based on subjects weight.
  Arms: Placebo
Biological: 1 mg/kg every 2 weeks — Subjects will receive placebo or active treatment every 2 weeks for a total of 9 doses. Duration of IV infusion is 60 minutes. Total dose is based on subjects weight.
  Arms: RN316: 1 mg/kg every 2 weeks
Biological: 2 mg/kg every 4 weeks — Subjects will receive placebo or active treatment every 2 weeks for a total of 9 doses. Duration of IV infusion is 60 minutes. Total dose is based on subjects weight.
  Arms: RN316: 2 mg/kg every 4 weeks
Biological: 4 mg/kg every 4 weeks — Subjects will receive placebo or active treatment every 2 weeks for a total of 9 doses. Duration of IV infusion is 60 minutes. Total dose is based on subjects weight.
  Arms: RN316: 4 mg/kg every 4 weeks
Biological: 4 mg/kg every 8 weeks — Subjects will receive placebo or active treatment every 2 weeks for a total of 9 doses. Duration of IV infusion is 60 minutes. Total dose is based on subjects weight.
  Arms: RN316: 4 mg/kg every 8 weeks
Biological: 8 mg/kg every 8 weeks — Subjects will receive placebo or active treatment every 2 weeks for a total of 9 doses. Duration of IV infusion is 60 minutes. Total dose is based on subjects weight.
  Arms: RN316: 8 mg/kg every 8 weeks
Biological: 12 mg/kg every 8 weeks — Subjects will receive placebo or active treatment every 2 weeks for a total of 9 doses. Duration of IV infusion is 60 minutes. Total dose is based on subjects weight.
  Arms: RN316: 12 mg/kg every 8 weeks

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of repeated doses of RN316 in eligible healthy volunteers. RN316 is an investigational drug that is currently being studied as a cholesterol lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* LDL-C must be greater or equal to 130 mg/dl
* BMI must be between 18.5 and 40 kg/m2

Exclusion Criteria:

* History of cardiovascular or cerebrovascular event during the past year.
* Poorly controlled type 1 or type 2 diabetes mellitus
* Subjects who have taken lipid lowering therapies within the last 3 months of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting or intolerable treatment related adverse events (AEs). | Every Scheduled Visit
Incidence, severity and causal relationship of treatment emergent AEs (TEAEs). | Every Scheduled Visit
Incidence of abnormal and clinically relevant safety laboratories. | Screening and Days 29, 57, 85, 113, 135, 141, 169 and 197
Abnormal and clinically relevant changes in vital signs, BP, and ECG parameters. | Every Scheduled Visit
Incidence of anti-drug-antibodies. | Baseline and Day 15 and monthly thereafter

SECONDARY OUTCOMES:
PK parameter estimates including but not be limited to: AUC, Tmax, Cmax terminal elimination half life (t1/2), Clearance (CL), volume of distribution at steady state (Vss), and accumulation ratio (R) of RN316. | Day 1 and every scheduled visit thereafter
Absolute and percentage change in LDL C from baseline. | Every scheduled visit except Day 1
Proportion of subjects who achieve a target LDL C of <100 mg/mL. | Every scheduled visit except Day 1
Proportion of subjects who achieve a target LDL C of <70 mg/dL. | Every scheduled visit except Day 1
Proportion of subjects achieving 50% decrease in LDL C from baseline. | Every scheduled visit except Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481002&StudyName=Multiple-Dose%20Safety%20Study%20Of%20RN316%20For%20TheTreatment%20Of%20Hypercholesterolemia